CLINICAL TRIAL: NCT03054636
Title: Short-term 2D Perfusion Angiography Pilot Study
Brief Title: Short-term Perfusion Angiography Pilot Study (SPA)
Acronym: SPA
Status: Terminated | Type: Observational
Why Stopped: After data review of enrolled pts, it was determined that initial study objectives would not be met w/ continuation of enrollment
Sponsor: Volcano Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 160201
Record Dates: First submitted 2017-02-13; First posted 2017-02-15 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The Short term Perfusion Angiography (SPA) study is designed to collect 2D Perfusion data from Critical Limb Ischemia (CLI) endovascular (interventional) procedures for information on device performance in a real-world setting.

DETAILED DESCRIPTION:
This clinical study is designed to collect pre and post procedural imaging data using 2D Perfusion (2DP) software in patients receiving an endovascular intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 years of age.
2. Subject or their legally authorized representative understands the research nature of the study and is willing and capable of providing informed consent
3. Subject has appropriate femoral arterial access
4. Subject presents with a Rutherford classification of 4 to 6.
5. Planned DSA with endovascular intervention below the knee on one or both limbs. This may include patients who undergo:

   1. Above the knee (ATK) and below the knee (BTK) intervention during the same procedure.
   2. Only BTK intervention.
   3. ATK intervention with staged future BTK intervention within 6 weeks of the initial procedure.

Exclusion Criteria:

1. Subjects whose ATK intervention is limited to only the common femoral or iliac arteries
2. Subject is unwilling or unable to comply with the protocol including all follow-up visits
3. Subject with active atrial fibrillation at time of procedure
4. Critical limb ischemia due to acute arterial occlusion.
5. Subject with documented ejection fraction < 40% and/or prolonged bradycardia (< 60 beats per minute)
6. Inability to collect toe pressure on index limb from subject
7. Subjects with history of or known reaction or sensitivity to contrast agent that cannot be pre-medicated or any other condition that precludes an endovascular intervention and DSA
8. Female subject of childbearing potential who is pregnant (she must have negative pregnancy test within the 48 hours prior to enrollment), or plans a pregnancy during study period,
9. Subject life expectancy < 3 months,
10. Subject is participating in a potentially confounding device or drug clinical trial that interferes with this study
11. Investigator considers subject to be a poor candidate for the study or believes that the patient may compromise the study, e.g., concomitant conditions (reasons will be documented) )

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 132 patients with critical limb ischemia (Rutherford classification 4, 5 or 6) considered candidates for a diagnostic angiogram and likely endovascular intervention expected to be enrolled into the SPA Study
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2017-01; Primary Completion 2019-02-14 (Actual); Study Completion 2019-02-14 (Actual)

PRIMARY OUTCOMES:
Safety (Freedom from Major Adverse Device Effects) | 30 days
  Freedom from Major Adverse Device Effects through 30 day visit.

CONTACTS AND LOCATIONS:
Overall Officials: Jihad Mustapha, MD, Principal Investigator — Metro Health Hospital; Larry J Diaz-Sandoval, MD, Principal Investigator — Metro Health Hospital
Locations (4):
- United States (4):
  - Miami Cardiac and Vascular Institute, Miami, Florida
  - Metro Health Hospital, Wyoming, Michigan
  - North Carolina Heart and Vascular, Raleigh, North Carolina
  - University Hospitals, Cleveland, Ohio